CLINICAL TRIAL: NCT04518150
Title: Clinical Outcomes of Combined Bilateral Uterine Artery Ligation and Bakri Balloon Tamponade During Cesarean Section in Patients With Placenta Previa: a Randomized Controlled Trial
Brief Title: Combined Bilateral Uterine Artery Ligation and Bakri Balloon During Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: aswu/270/9/18
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Trial
Who Masked: Participant
Masking Description: single blind randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): patients with placenta previa undergoing cesarean section underwent bilateral uterine artery ligation plus insertion of Bakri balloon
  Interventions: Device: Bakri balloon; Procedure: Bilateral Uterine Artery Ligation
- control group (Active Comparator): patients with placenta previa undergoing cesarean section underwent insertion of Bakri balloon
  Interventions: Device: Bakri balloon

INTERVENTIONS:
Device: Bakri balloon — the Bakri balloon was inserted into the lower uterine segment through the uterine incision by passing the balloon shaft through the cervix with an assistant pulling vaginally
  Other Names: BBT
Procedure: Bilateral Uterine Artery Ligation — The peritoneum over the vesico-uterine pouch already being incised horizontally, the peritoneum over the uterine isthmus and cervix was dissected downwards, and this dissection was then extended laterally.
  Other Names: BUAL
  Arms: study group

SUMMARY:
This study will be performed to compare the effectiveness of routine Bakri balloon tamponade and Bilateral Uterine Artery Ligation during cesarean section in patients with placenta previa

DETAILED DESCRIPTION:
Intraoperative methods to control profuse bleeding during cesarean section in patients with placenta previa include uterine packing, balloon tamponade, uterine compression sutures, arterial ligation, uterine artery embolization, and hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing elective cesarean delivery for complete placenta previa which not respond uterotonic and simple hemostatic maneuvers like placental bed hemostatic sutures

Exclusion Criteria:

* patients with the high possibility of morbid adherent placenta
* those presented with severe antepartum hemorrhage
* Patients with cardiac, hepatic, renal, or thromboembolic disease;
* patient refuses to consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women undergoing elective cesarean delivery for complete placenta previa which not respond uterotonic and simple hemostatic maneuvers like placental bed hemostatic sutures
Enrollment: 150 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
mean Blood loss after placental separation | 30 minutes
  by using weight of soaked towels (weight of soaked towel - weight of dry towel) and amount of blood in suction set

SECONDARY OUTCOMES:
The number of participant needed for blood transfusion | 24 hours
  Calculation of the number of participant needed for blood transfusion
Number of Participants with postpartum hemorrhage | 24 hours
  number pf participants with blood loss > 1000ml

CONTACTS AND LOCATIONS:
Overall Officials: nahla w Shady, md, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No